CLINICAL TRIAL: NCT01374022
Title: Randomized Controlled Trial of Maximum Alveolar Recruitment Maneuver Plus Titrated PEEP Versus ARDSNet Strategy for ARDS
Brief Title: ART - Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial
Acronym: ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE - 0025.1.160.000-11
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Respiratory Distress Syndrome, Adult; Randomized Controlled Trial; Respiration, Artificial
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ART Strategy (Experimental): maximum alveolar recruitment plus PEEP titration
  Interventions: Other: ART Strategy
- ARDSNet Strategy (Active Comparator): standard strategy (ARDSNet)
  Interventions: Other: ARDSNet Strategy

INTERVENTIONS:
Other: ART Strategy — Maximum alveolar recruitment maneuver in association with PEEP titrated by the static compliance of respiratory system.
  Arms: ART Strategy
Other: ARDSNet Strategy — Conventional mechanical ventilation strategy.
  Arms: ARDSNet Strategy

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a common scenario in intensive care unit. Discussions about it is exponentially growing up due its high mortality rates all over the world and low quality of life among survivors. Mechanical ventilation is recognized to play an important role in treatment of patients with ARDS. However, mechanical ventilation itself has the potential to produce or worsen alveolar injury if inadequate strategies are chosen. Several studies compared different mechanical ventilation strategies in ARDS but the results remain uncertain regarding their influence on survival in patients with ARDS. Thus, this is a multicentric randomized controlled trial, with allocation concealment and intention to treat analysis to investigate if maximum alveolar recruitment maneuver in association to Positive end-expiratory pressure (PEEP) titrated by static compliance of respiratory system (ART strategy) is able to increase 28 days survival in patients with moderate to severe ARDS compared to conventional strategy proposed by the ARDS Clinical Network (ARDSNet strategy). Patients considered to this trial are those in mechanical ventilation with diagnosis of moderate to severe ARDS less than 72hours. Patients included will be randomized to receive ART strategy or ARDSNet strategy and will be followed until hospital discharge, 28 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* intubated, mechanically ventilated patients with diagnosis of moderate to severe ARDS less than 72 hours

Exclusion Criteria:

* age less than 18 years
* use of vasopressor drugs in increasing doses over the last 2 hours or mean arterial blood pressure less than 65mmHg
* presence of any contraindication to hypercapnia as intracranial hypertension or acute coronary syndrome
* pneumothorax, pneumomediastinum, subcutaneous emphysema or pneumatocele
* patient with no therapeutic perspective, candidates for palliative care exclusively
* patient previously randomized in the ART

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Survival in 28 days | 28 days
  Survival within 28 days from randomization

SECONDARY OUTCOMES:
Lenght of ICU stay | Maximum 6-months
  Length of hospital stay from randomization to ICU discharge
Lenght of hospital stay | Maximum 6 months
  Length of hospital stay from randomization to hospital discharge
Pneumothorax requiring drainage | 7 days
  We consider as pneumothorax requiring chest tube within 7 days any case that is possibly due to barotrauma, that is, we do not consider cases judged to be clearly caused by invasive procedures such as central venous punction or thoracocentesis.
Barotrauma | 7 days
  We consider as barotrauma within 7 days any pneumothorax, pneumomediastinum, subcutaneous emphysema or pneumatocele > 2cm detected on image exams between randomization and 7 days, except those judged to be clearly caused by invasive procedures.
Days free of mechanical ventilation | 28 days
  Number of days alive and out of mechanical ventilation between randomization and 28 days after randomization.
ICU survival | Maximum 6-months
  Survival at ICU discharge.
In-hospital survival | Maximum 6-months
  Survival at hospital discharge.
6-month survival | 6 months
  Survival within 6 months after randomization

OTHER OUTCOMES:
Need of commencement/increase of vasopressors or hypotension (MAP < 65mmHg) in the first hour; | 1 hour
  Need of commencement/increase of vasopressors or hypotension (MAP < 65mmHg) in the first hour after randomization.
Hypoxemia (PaO2 < 55mmHg) in the first hour | 1 hour
  Hypoxemia (PaO2 < 55mmHg) in the first hour after randomization
Severe acidosis (pH < 7.10) in the first hour | 1 hour
  Severe acidosis (pH < 7.10) in the first hour after randomization
Cardiorespiratory arrest within 24 hours | 24 hours
  Cardiorespiratory arrest defined as unexpected cardiac arrest, not due to progressive refractory shock within 24 hours after randomization.
Deaths with refractory hypoxemia within 7 days | 7 days
  Death with refractory hypoxemia, defined as PaO2 < 55 mmHg in the last arterial blood gas analysis with FiO2 = 100%.
Death with refractory acidosis within 7 days | 7 days
  Death with refractory acidosis within 7 days, defined as pH ≤ 7.10 in the last arterial blood gas analysis
Death with barotrauma within 7 days | 7 days
  Death with barotrauma within 7 days after randomization. We consider as barotrauma any pneumothorax, pneumomediastinum, subcutaneous emphysema or pneumatocele > 2cm detected on image exams, except those judged to be clearly caused by invasive procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, PhD, Principal Investigator — Hospital do Coracao; Carlos RR Carvalho, MD, PhD, Study Chair — Hospital do Coracao, Faculdade de Medicina da Universidade de Sao Paulo
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Zampieri FG, Costa EL, Iwashyna TJ, Carvalho CRR, Damiani LP, Taniguchi LU, Amato MBP, Cavalcanti AB; Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial Investigators. Heterogeneous effects of alveolar recruitment in acute respiratory distress syndrome: a machine learning reanalysis of the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial. Br J Anaesth. 2019 Jul;123(1):88-95. doi: 10.1016/j.bja.2019.02.026. Epub 2019 Apr 5. PMID 30961913
- [Derived] Damiani LP, Berwanger O, Paisani D, Laranjeira LN, Suzumura EA, Amato MBP, Carvalho CRR, Cavalcanti AB. Statistical analysis plan for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART). A randomized controlled trial. Rev Bras Ter Intensiva. 2017 Apr-Jun;29(2):142-153. doi: 10.5935/0103-507X.20170024. PMID 28977255
- [Derived] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Derived] Morais CC, De Santis Santiago RR, Filho JR, Hirota AS, Pacce PH, Ferreira JC, Camargo ED, Amato MB, Costa EL. Monitoring of Pneumothorax Appearance with Electrical Impedance Tomography during Recruitment Maneuvers. Am J Respir Crit Care Med. 2017 Apr 15;195(8):1070-1073. doi: 10.1164/rccm.201609-1780LE. No abstract available. PMID 28409685
- [Derived] ART Investigators. Rationale, study design, and analysis plan of the Alveolar Recruitment for ARDS Trial (ART): study protocol for a randomized controlled trial. Trials. 2012 Aug 28;13:153. doi: 10.1186/1745-6215-13-153. PMID 22929542